CLINICAL TRIAL: NCT04486170
Title: Assessment of Patient Education as a Method of Optimizing Postpartum Care in Women With Hypertension
Brief Title: Assessment of Postpartum Education to Improve Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB STUDY 00001865
Record Dates: First submitted 2020-07-08; First posted 2020-07-24 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Hypertension in Pregnancy; Postpartum Preeclampsia
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: Current hospital education practices (No Intervention): The control group will receive standard of care postpartum educational materials provided by the nursing and resident physician staff. The will be asked to complete a brief questionnaire to determine if they would be interested in receiving education in a video formal.
- Intervention group: Standardized video and pamphlet (Experimental): The subjects enrolled in the invention group will be shown a 5 minute educational video on hypertension in the postpartum period. The patients will be shown the video on the ipad while they are in the comfort of their room. They will also be provided with a pamphlet with similar information that was discussed in the video. They will also be asked to complete a brief, anonymous survey to assess patient satisfaction with the video shown, no patient identifiers will be collected.
  Interventions: Other: Education provided via a video format

INTERVENTIONS:
Other: Education provided via a video format — The intervention group will be shown a 5 minute educational video on hypertension in the postpartum period. The patients will be shown the video on the ipad while they are in the comfort of their room and the investigator will step outside. At the conclusion of the video, the investigator will return into the patient room and provide a pamphlet with similar information that was discussed in the video for them to take home.
  Other Names: Education provided in a pamphlet
  Arms: Intervention group: Standardized video and pamphlet

SUMMARY:
This is a prospective single centered randomized control study for postpartum patients diagnosed with hypertension. Participants that meet inclusion criteria will be approached while they are inpatient. After enrollment, all study subjects will receive an automated blood pressure cuff and instructions on how to use it. Study participants in the intervention group will be provided with educational material. The investigators hypothesize education in postpartum women with hypertension can improve patient compliance with attendance at postpartum care appointments.

DETAILED DESCRIPTION:
The study group: postpartum women with a diagnosis of either chronic hypertension, gestational hypertension, preeclampsia without severe features, preeclampsia with severe features, chronic hypertension with superimposed preeclampsia with and without severe features.

Recruitment: postpartum patients that meet the inclusion criteria will be approached postpartum while they are still hospitalized. Once the study subjects are enrolled, they will receive the same automatic blood pressure cuff and basic teaching on how to use it. All study subjects will be asked to check their blood pressure once a day. The study subjects will be advised that if systolic blood pressure is > 160 or the diastolic blood pressure >110, the study subjects are asked to remain seated and repeat the BP measurement in 15 minutes, if still elevated the study subject will be advised to call labor and delivery or proceed to labor and delivery triage for further evaluation. All study subjects will be asked to follow up for a blood pressure check 3-10 days after discharge home. All study subjects will be weighed prior to discharge.

The study subject is then randomized to the control or intervention group. Both groups will receive a survey. After the intervention group undergoes the educational component, this will be the last time the study subjects meet with the investigator.

The data will be collected on an excel spreadsheet. Patient identifiers will be removed once the study is completed. However, de-identified data may be used for future studies. The database will be password protected on an excel spreadsheet and secured behind the Medstar Washington Hospital Center firewall computers. Access to these databases is restricted to the PI and the co-investigators. The data will be statistically analyzed in order to answer the primary and secondary outcomes.

Power analysis: At Washington hospital center, the current attendance within 10 day postpartum follow up appointments is 40% and at the 6 week appointment it is 70%. Based on this data the investigator wants to evaluate if this postpartum education intervention can cause a 100% difference in attendance within 10 days postpartum: 40% attendance which is the current attendance rate (control) versus 80% (goal for the intervention group): enrollment of 46 patients is required.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum with diagnosis of Hypertension is defined as chronic hypertension, gestational hypertension, preeclampsia without severe features, preeclampsia with severe features, chronic hypertension with superimposed preeclampsia with and without severe features.
* At least 18 years or older
* English speaking patient and also able to read in English
* Plan to receive postpartum care at Washington Hospital Center

Exclusion Criteria:

* Women who do not intend to follow up at Washington Hospital Center
* Suffered from intrauterine fetal demise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Compliance with postpartum care | This outcome will be evaluated within 10 days of discharge
  The investigators will perform a retrospective chart review to determine if the study participant attended the postpartum BP check appointment
Compliance with postpartum care | This outcome will be evaluated within 6 weeks of delivery
  The investigators will perform a retrospective chart review to determine if the study participant attended the postpartum BP check appointment

SECONDARY OUTCOMES:
Incidence of postpartum re-admission for hypertension related concerns | This outcome will be evaluated within 6 weeks of delivery
  The investigators will retrospectively review if the study participants are re-admitted for hypertension related concerns
Incidence of postpartum labor and delivery triage visits | This outcome will be evaluated within 6 weeks of delivery
  The investigators will retrospectively review if the study participants are evaluated in the labor and delivery triage for hypertension related concerns
Incidence of postpartum emergency department visits | This outcome will be evaluated within 6 weeks of delivery
  The investigators will retrospectively review if the study participants are evaluated in the emergency department for hypertension related concerns
Evaluate weight (kg) change | This outcome will be evaluated upon hospital admission
  The investigators will retrospectively compare the participants weight upon delivery admission to weight upon discharge and within 6 weeks of delivery
Evaluate weight (kg) change | This outcome will be evaluated upon hospital discharge
  The investigators will retrospectively compare the participants weight upon delivery admission to weight upon discharge and within 6 weeks of delivery
Evaluate weight (kg) change | This outcome will be evaluated within 6 week after delivery
  The investigators will retrospectively compare the participants weight upon delivery admission to weight upon discharge and within 6 weeks of delivery
Incidence of stroke | This outcome will be evaluated within 6 weeks of delivery
  The investigators will retrospectively review if the study participant suffered a stroke
Incidence of maternal death | This outcome will be evaluated within 6 weeks of delivery
  The investigators will retrospectively review maternal death during this study period
Participant satisfaction with postpartum education using likert scale | This outcome will be evaluated at time of recruitment, within 48hours
  A likert scale survey will be administered by the investigator to the intervention and control group, the satisfaction score will be compared between both groups. The scale is reported as follows: 1 (Strongly disagree) 2 3 (neutral) 4 5 (strongly agree).
Participant satisfaction with postpartum education | This outcome will be evaluated at time of recruitment, within 48hours
  A survey will be administered by the investigator to the intervention and control group, the satisfaction score will be compared between both groups. The responses are either Yes or No. For most questions, answering yes would be a favorable response.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Iqbal, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No